CLINICAL TRIAL: NCT04074551
Title: A Randomized, Double-blinded, Multi-center, Phase III Study to Compare The Efficacy and Safety of Co-administered HGP0608, HGP0904 and HCP1306 Versus HCP1701 in Patients With Hypertension and Dyslipidemia
Brief Title: A Phase 3 Study to Compare the Efficacy and Safety of Co-administered HGP0608, HGP0904 and HCP1306 Versus HCP1701 in Patients With Hypertension and Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-AMOS-301
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Losartan; Amlodipine; Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): HCP1701
  Interventions: Drug: HCP1701
- Active Comparator 1 (Active Comparator): HGP0904, HGP0608
  Interventions: Drug: Losartan; Drug: Amlodipine
- Active Comparator 2 (Active Comparator): HGP0608, HCP1306
  Interventions: Drug: Losartan; Drug: Rosuvastatin and Ezetimibe

INTERVENTIONS:
Drug: HCP1701 — HCP1701
  Arms: Experimental
Drug: Losartan — Losartan
  Arms: Active Comparator 1; Active Comparator 2
Drug: Amlodipine — Amlodipine
  Arms: Active Comparator 1
Drug: Rosuvastatin and Ezetimibe — Rosuvastatin and Ezetimibe
  Arms: Active Comparator 2

SUMMARY:
A Randomized, Double-blinded, Multi-center, Phase III Study to Compare The Efficacy and Safety of Co-administered HGP0608, HGP0904 and HCP1306 versus HCP1701 in Patients with Hypertension and Dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19
* Patients who understood the contents and purpose of this trial and signed informed consent form
* Patients with essential hypertension and dyslipidemia

Exclusion Criteria:

* Patients with differences between arms greater than 20 mmHg for mean sitSBP or 10 mmHg for mean sitDBP
* Patients with mean sitSBP ≥ 180 mmHg or mean sitDBP ≥ 110 mmHg
* Concomitant administration of cyclosporine
* Tolerance or Hypersensitivity Angiotensin II receptor blocker or HMG-CoA reductase inhibitor, Calcium channel blocker(dihydropyridine) or Multi-drug allergy
* Hereditary angioedema or medical history of angioedema in the treatment of ACE inhibitors or angiotensin II receptor blockers
* Fibromyalgia, myopathy, rhabdomyolysis or acute myopathy or medical history of adverse effect to statin
* CPK normal range > 2 times
* Secondary hypertension and suspected secondary hypertension
* Orthostatic hypotension with symptoms
* Uncontrolled primary hypothyroidism(TSH normal range ≥ 1.5 times)
* Severe hepatopathy or active hepatopathy (AST or ALT normal range ≥ 3 times)
* Active gout or hyperuricemia(uric acid ≥ 9mg/dL)
* IDDM or uncontrolled type 2 diabetes mellitus (HbA1c > 9%)
* Ventricular arrhythmia
* Medical history

  * Severe heart disease(heart failure of NYHA class III-IV)
  * Severe cerebrovascular disease within 6 months (cerebral infarction, cerebral hemorrhage), hypertensive encephalopathy, transient cerebral ischemic attack(TIA)
  * Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant stenosis in aortic valve or mitral valve
  * Ischemic heart disease(myocardial infarction, angina) within 6months
  * Angioplasty or coronary artery bypass graft(CABG) surgery within 6months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in LDL-C (%) | baseline, 8 weeks
  Experimental, Active Control 1
Change from baseline in sitting systolic blood pressure | baseline, 8 weeks
  Experimental, Active Control 2

SECONDARY OUTCOMES:
Change from baseline in LDL-C (%) | baseline, 8 weeks
  Experimental, Active Control 2
Change from baseline in sitting systolic blood pressure | baseline, 8 weeks
  Experimental, Active Control 1
Change from baseline in LDL-C (%) | baseline, 4 weeks
Change from baseline in sitting systolic blood pressure | baseline, 4 weeks
Change from baseline in TC, HDL-C, TG (%) | baseline, 4 weeks, 8 weeks
Change from baseline in sitting distolic blood pressure | baseline, 4 weeks, 8 weeks
Proportion of subject achieving LDL-C control | baseline, 4 weeks, 8 weeks
Proportion of subjects achieving blood pressure control | baseline, 4 weeks, 8 weeks
Proportion of responder for blood pressure | baseline, 4 weeks, 8 weeks
Proportion of subject achieving both LDL-C and blood pressure control | baseline, 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim MC, Ahn Y, Kim MH, Kim SY, Hong TJ, Rhee MY, Kim SH, Hong SJ, Kim H, Kim W, Chae IH, Kang DH, Kim BK, Kim HS. A Randomized, Multicenter, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of a Quadruple Combination of Amlodipine, Losartan, Rosuvastatin, and Ezetimibe in Patients with Concomitant Essential Hypertension and Dyslipidemia. Am J Cardiovasc Drugs. 2023 Jul;23(4):441-454. doi: 10.1007/s40256-023-00590-9. Epub 2023 Jul 3. PMID 37395974